CLINICAL TRIAL: NCT02708524
Title: Clinical Study of Approved and Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5808
Record Dates: First submitted 2016-03-03; First posted 2016-03-15 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Senofilcon C Wearers (Experimental): Senofilcon C Wearers will wear the Senofilcon C Contact Lenses as daily wear for 30 (-2/+6) days.
  Interventions: Device: Senofilcon C Contact Lens
- Comfilcon A Wearers (Active Comparator): Comfilcon A Wearers will wear the Comfilcon A Contact Lens as daily wear for 30 (-2/+6) days.
  Interventions: Device: Comfilcon A Contact Lens
- Lotrafilcon B Wearers (Active Comparator): Lotrafilcon B Wearers will wear the Lotrafilcon B Contact Lens as daily wear for 30 (-2/+6) days.
  Interventions: Device: Lotrafilcon B Contact Lens
- Samfilcon A Wearers (Active Comparator): Samfilcon A Wearers will wear the Samfilcon A Contact Lens as daily wear for 30 (-2/+6) days.
  Interventions: Device: Samfilcon A Contact Lens

INTERVENTIONS:
Device: Senofilcon C Contact Lens
  Other Names: senofilcon C
  Arms: Senofilcon C Wearers
Device: Comfilcon A Contact Lens
  Other Names: comfilcon A
  Arms: Comfilcon A Wearers
Device: Lotrafilcon B Contact Lens
  Other Names: lotrafilcon B
  Arms: Lotrafilcon B Wearers
Device: Samfilcon A Contact Lens
  Other Names: samfilcon A
  Arms: Samfilcon A Wearers

SUMMARY:
This is a multi-site, 5-visit, double-masked, dispensing study comparing an investigational contact lens with currently-marketed contact lenses. The objective of the study is to evaluate the comfort of the lenses when worn for 30 (-2/+6) days on daily wear modality.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 18 to 40 years of age at the time of consent.
4. The subject's spherical equivalent distance refraction must be in the range of -1.25 to -6.00 in each eye.
5. The subject's refractive cylinder must be ≤1.00D in each eye.
6. The subject must have best corrected visual acuity of 20/30 or better in each eye.
7. The subject must be a habitual frequent replacement (reusable) daily wear spherical silicone hydrogel soft contact lens wearer in both eyes.
8. The subject must be able to wear contact lenses for a minimum of 8 hours, 4 days per week.
9. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Any known sensitive/allergic to Ingredients of OPTI-FREE® PureMoist® solution.
5. Any daily disposable, extended wear, monovision, toric or multi-focal contact lens correction.
6. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
7. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
8. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
9. Any ocular infection.
10. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
11. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
12. History of binocular vision abnormality or strabismus.
13. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV), by self-report).
14. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Montgomery, Alabama
  - Fruit Cove, Florida
  - Jacksonville, Florida
  - Longwood, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Roswell, Georgia
  - Bloomington, Illinois
  - East Lansing, Michigan
  - Medina, Minnesota
  - Closter, New Jersey
  - Vestal, New York
  - Granville, Ohio
  - Jacksonville, Texas
  - Salt Lake City, Utah
  - Roanoke, Virginia
  - West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 554 subjects were enrolled in this study. Of the enrolled subjects 6 subjects did not meet the eligibility criteria and 548 subjects were dispensed a study lens. Of the dispensed subjects 535 subjects completed the study and 13 subjects were discontinued.
Groups:
- Senofilcon C: Subjects that were randomized to receive the senofilcon C lens throughout the duration of the study.
- Comfilcon A: Subjects that were randomized to receive the comfilcon A lens throughout the duration of the study.
- Lotrafilcon B: Subjects that were randomized to receive the lotrafilcon B lens throughout the duration of the study.
- Samfilcon A: Subjects that were randomized to receive the samfilcon A lens throughout the duration of the study.
Period: Overall Study
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Started | 139 | 136 | 137 | 136
Completed | 135 | 130 | 134 | 136
Not Completed | 4 | 6 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lens Discomfort | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Dispensed incorrect study lens | 0 | 1 | 1 | 0
Not completed — Did not wear lens at final visit | 0 | 1 | 0 | 0
Not completed — Subject lost study lens | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Senofilcon C: All subjects that wore the senofilcon C lens throughout the duration of the study.
- Comfilcon A: All subjects that wore the comfilcon A lens throughout the duration of the study.
- Lotrafilcon B: All subjects that wore the lotrafilcon B lens throughout the duration of the study.
- Samfilcon A: All subjects that wore the samfilcon A lens throughout the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A | Total
Number analyzed (Participants) | 139 | 136 | 137 | 136 | 548
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (6.24) | 27.7 (5.86) | 28.6 (5.63) | 28.8 (6.56) | 28.6 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 98 | 86 | 92 | 364
  Male | 51 | 38 | 51 | 44 | 184
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 2 | 6 | 10 | 20
  Black or African American | 13 | 10 | 9 | 12 | 44
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  White | 119 | 122 | 122 | 113 | 476
  Other | 3 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 139 | 136 | 137 | 136 | 548

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort Composite Score
Description: Subjective Overall Comfort was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.Range is 0 to 120. CLUE was collect at Baseline, Post Lens Fit 1-, 2-, 3- and 4- week follow-ups.
Time Frame: Up to 1 month Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: average clue score
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
average clue score
  Baseline | 65.17 (23.612) | 68.58 (21.993) | 66.45 (22.864) | 65.46 (22.220)
  Post Fit | 66.65 (16.198) | 62.11 (18.814) | 52.27 (22.762) | 64.40 (19.305)
  1-Week Follow-up | 67.29 (22.863) | 55.78 (26.628) | 54.40 (26.260) | 56.96 (25.508)
  2-Week Follow-up | 64.18 (22.455) | 55.56 (24.955) | 53.09 (26.908) | 55.01 (24.817)
  3-Week Follow-up | 61.31 (23.850) | 55.01 (27.069) | 52.17 (26.585) | 53.72 (26.794)
  4-Week Follow-up | 60.74 (26.121) | 56.32 (27.549) | 51.15 (28.609) | 52.61 (27.549)

2. Primary Outcome: Overall Comfort Individual Item
Description: Overall Comfort was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Responses are on a 5 likert scale (Excellent, Very Good, Good, Fair and Poor). Only the percentage of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: 1 month follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 78 | 82 | 80 | 77
  1-Week Follow-up | 79.1 | 50.7 | 51.9 | 56.6
  2-Week Follow-up | 70.9 | 54.7 | 48.2 | 54.5
  3-Week Follow-up | 69.4 | 50 | 45.2 | 53
  4-Week Follow-up | 68.7 | 54.6 | 46.2 | 50

3. Primary Outcome: Comfort at the End of the Day Individual Item
Description: Comfort at the End of the Day was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are on a 5 like-rt scale (Excellent, Very Good, Good, Fair and Poor). Only the percentage of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 57.5 | 64.6 | 60.9 | 64.0
  1-Week Follow-up | 64.2 | 47.0 | 43.6 | 49.3
  2-Week Follow-up | 59.0 | 48.4 | 45.9 | 49.3
  3-Week Follow-up | 52.2 | 42.3 | 42.1 | 45.6
  4-Week Follow-up | 55.2 | 43.0 | 39.8 | 45.6

4. Primary Outcome: Comfort Each and Everyday Individual Item
Description: Comfort each and everyday was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are on a 5 likert scale (Excellent, Very Good, Good, Fair and Poor). Only the percentage of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 73.2 | 76.1 | 78.3 | 76.5
  1-Week Follow-up | 79.1 | 59.2 | 54.2 | 56.6
  2-Week Follow-up | 70.9 | 58.5 | 52.6 | 53.0
  3-Week Follow-up | 70.9 | 54.6 | 48.2 | 53.0
  4-Week Follow-up | 68.7 | 54.6 | 48.9 | 52.2

5. Primary Outcome: Frequency of Lens Awareness Individual Item
Description: Frequency of Lens Awareness was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are scaled as (Always, Frequently, Occasionally, Rarely, Never or Don't Know). Only the number of participants that reported Rarely or Never (Top-Two-Box) was reported here.
Time Frame: 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 73.2 | 74.5 | 77.4 | 75.8
  1-Week Follow-up | 75.4 | 61.6 | 54.9 | 66.2
  2-Week Follow-up | 78.3 | 63.9 | 45.6 | 66.2
  3-Week Follow-up | 73.2 | 60.0 | 54.2 | 59.6
  4-Week Follow-up | 75.4 | 60 | 51.2 | 63.2

6. Primary Outcome: Frequency of Experiencing Dryness Individual Item
Description: Frequency of Experiencing Dryness was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are scaled as (Always, Frequently, Occasionally, Rarely, Never or Don't Know). Only the number of participants that reported Rarely or Never (Top-Two-Box) was reported here.
Time Frame: 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 62.7 | 67.7 | 71.4 | 67.6
  1-Week Follow-up | 67.9 | 62.5 | 53.4 | 62.5
  2-Week Follow-up | 67.2 | 50.1 | 50.4 | 59.6
  3-Week Follow-up | 64.2 | 59.2 | 51.2 | 56.6
  4-Week Follow-up | 68.0 | 55.4 | 50.4 | 55.9

7. Primary Outcome: Making Your Eyes Feel Moist Throughout the Day Individual Item
Description: Making your eyes feel moist throughout the day was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are on a 5 likert scale (Excellent, Very Good, Good, Fair and Poor). Only the percentage of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: Up to 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 68.6 | 52.3 | 43.7 | 55.2
  1-Week Follow-up | 58.6 | 52.3 | 43.7 | 55.2
  2-Week Follow-up | 58.2 | 53.1 | 49.7 | 50.0
  3-Week Follow-up | 61.2 | 48.5 | 45.9 | 48.6
  4-Week Follow-up | 64.9 | 54.6 | 43.6 | 49.3

8. Secondary Outcome: Subjective Overall Quality of Vision Composite Score
Description: Subjective Overall Quality of Vision was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. CLUE was collect at Baseline, Post Lens Fit 1-, 2-, 3- and 4- week follow-ups.
Time Frame: Up to 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
units on a scale
  Baseline | 63.79 (20.515) | 63.31 (20.510) | 64.12 (19.822) | 62.34 (19.383)
  Post Fit | 69.45 (14.896) | 68.96 (16.272) | 65.58 (17.300) | 67.07 (16.741)
  1- Week Follow-up | 62.32 (20.897) | 63.55 (20.586) | 59.36 (22.076) | 58.61 (19.359)
  2- Week Follow-up | 64.77 (20.222) | 61.66 (20.504) | 58.29 (23.543) | 56.54 (21.679)
  3- Week Follow-up | 63.22 (21.125) | 61.41 (22.137) | 57.27 (22.463) | 53.65 (22.128)
  4- Week Follow-up | 63.30 (22.852) | 60.99 (22.573) | 56.63 (24.879) | 53.57 (23.100)

9. Secondary Outcome: Overall Quality of Vision Individual Item
Description: Overall Quality of Vision was assessed using a questionnaire item at Baseline, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are on a 5 likert scale (Excellent, Very Good, Good, Fair and Poor). Only the number of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: Up to 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Baseline | 82.9 | 86.9 | 91.0 | 84.5
  1- Week Follow-up | 89.5 | 77.7 | 74.9 | 78.7
  2- Week Follow-up | 82.8 | 77.7 | 69.1 | 71.3
  3- Week Follow-up | 83.6 | 76.9 | 69.9 | 66.9
  4- Week Follow-up | 85.1 | 76.2 | 63.2 | 61.0

10. Secondary Outcome: Overall Opinion Individual Item
Description: Overall Opinion was assessed using a questionnaire item at Post Fit, 1-week, 2-week, 3-week and 4-week follow-up. Reposes are on a 5 likert scale (Excellent, Very Good, Good, Fair and Poor). Only the percentage of participants that reported Excellent or Very good (Top-Two-Box) was reported here.
Time Frame: Up to 1 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Number analyzed (Participants) | 134 | 130 | 133 | 136
percentage of participants
  Post Fit | 85.8 | 73.8 | 60.9 | 80.9
  1- Week Follow-up | 75.4 | 49.3 | 42.1 | 54.5
  2- Week Follow-up | 66.5 | 47.7 | 42.1 | 47.8
  3- Week Follow-up | 62.7 | 43.9 | 42.9 | 39.7
  4- Week Follow-up | 59.0 | 43.9 | 38.3 | 41.1

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 month per subject.
Arm/Group | Senofilcon C | Comfilcon A | Lotrafilcon B | Samfilcon A
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/136 | 0/137 | 1/136
Other Adverse Events (participants affected / at risk) | 0/139 | 0/136 | 0/137 | 0/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon C (N=139) | Comfilcon A (N=136) | Lotrafilcon B (N=137) | Samfilcon A (N=136)
Muscle Spasm in Chest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to the study article.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days